CLINICAL TRIAL: NCT00264186
Title: Impact of rhCu/Zn SOD on Inflammation-Induced Impairment of Vascular Reactivity
Brief Title: Recombinant Human Superoxide Dismutase (rhSOD) and Vascular Reactivity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Polymun Scientific, Vienna, Austria (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: LPS-rhSOD
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation | interventions — Lipopolysaccharides; Floors and Floorcoverings; Nitroglycerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: LPS 2 ng/kg intravenous (IV) bolus
Drug: rhSOD 82,000 IU (8.2 mg)/min intraarterially
Drug: Norepinephrine 60, 120, 240 pmol/min intraarterially over 5 min/dose level (two times; pre-dose and +3.5 hrs)
Drug: Acetylcholine 6.25, 12.5, 25 nmol/min intraarterially over 3 min/dose level (two times; pre-dose and +3.5 hrs)
Drug: Glyceroltrinitrate (nitroglycerine) 4, 8, 16 nmol/min over 3 min/dose level (two times; pre-dose and +3.5 hrs)

SUMMARY:
Inflammation is characterised by an increased risk for cardiovascular events. Dysfunction of the vascular endothelium caused by oxidative stress might provide a mechanistic link. In acute and chronic inflammation, oxidative stress occurs when the production of reactive oxygen species [ROS] (including superoxide anions [O2-]) exceeds the capacity of the endogenous antioxidant defense systems, resulting in ROS-mediated damage. Recombinant human superoxide dismutase (rhSOD) has shown potent antioxidant properties in in-vitro and animal studies and has been tested in phase I clinical trials in humans. rhSOD could offer a therapeutic option for vascular dysfunction in diseases associated with increased oxidative stress. The investigators, therefore, want to test if the hyporesponsiveness to vasoactive drugs (norepinephrine, acetylcholine and glyceroltrinitrate) during acute inflammation by low-dose lipopolysaccharide (LPS) is due to the increased production of superoxide anions, which could be scavanged by the radical scavenger rhSOD.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 18 and 45 years
* Nonsmokers
* Body mass index between 15th and 85th percentile
* Normal findings in medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, or participation in a clinical trial in the 3 weeks preceding the study
* Evidence of hypertension, pathologic hyperglycemia, or hyperlipidemia
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks
* History of hypersensitivity to the trial drug or to drugs with a similar chemical structure

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43
Dates: Start 2005-06

PRIMARY OUTCOMES:
Forearm blood flow responses to acetylcholine, nitroglycerine and norepinephrine (ratio between intervention and control arm)

SECONDARY OUTCOMES:
Markers of inflammation and oxidative stress, change in MAP, change in pulse rate, subjective symptoms and body temperature; antibodies against rhSOD

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolzt, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna - General Hospital of the City of Vienna AKH, Vienna, Vienna, Austria